CLINICAL TRIAL: NCT01534234
Title: Clinical Trial of the SonRtip Lead and Automatic AV-VV Optimization Algorithm in the PARADYM RF SonR CRT-D
Acronym: RESPOND-CRT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MicroPort CRM (Industry)
Collaborators: Sorin CRM (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITSY06 - RESPOND CRT
Expanded Access: Available
Record Dates: First submitted 2011-09-27; First posted 2012-02-16 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure NYHA Class III and Ambulatory IV
Keywords: CRT-D device; Severe HF (NYHA Class III or ambulatory IV); stable, optimal drug regimen; sinus rhythm

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- SonR group (Experimental): SonR CRT Optimization
  Interventions: Device: PARADYM RF SONR
- ECHO group (Active Comparator): Echocardiographic Optimization
  Interventions: Device: PARADYM RF SONR

INTERVENTIONS:
Device: PARADYM RF SONR — SonR CRT Optimization
  Other Names: Automatic Hemodynamic CRT Optimization
  Arms: SonR group
Device: PARADYM RF SONR — Echocardiography Optimization
  Other Names: Echo Optimization
  Arms: ECHO group

SUMMARY:
The objective of this study is to assess the safety and effectiveness of the automatic atrioventricular (AV) delay and interventricular (VV) delay optimization algorithm used in the PARADYM RF SONR Cardiac Resynchronization Therapy with Defibrillation (CRT-D) device (Model 9770) in combination with the SonRtip Lead, which includes a SonR sensor in the tip of the atrial pacing lead, and compatible SmartView programming software.

This study will evaluate the effectiveness of the automatic optimization algorithm in increasing the rate of patients responding to the therapy as compared to an echocardiographic optimization method.

This study will also evaluate the safety and effectiveness of the SonRtip atrial pacing lead.

DETAILED DESCRIPTION:
Since the introduction of cardiac resynchronization therapy (CRT) on a large scale, it has been observed that approximately 30% of recipient patients are non-responsive to therapy. This non-responsiveness can be decreased by optimizing the device programming, particularly the stimulation rate, paced and sensed atrioventricular (AV) delay, and the interventricular (VV) delay.

All CRT patients need a 100% rate of ventricular capture, but beyond this the achievement of therapy effectiveness requires the identification of the optimal pacing configuration, which varies among patients. The optimization of CRT systems, usually based on ultrasound imaging is time-consuming and the number of patients in need of multiple optimization procedures due to ventricular remodeling is growing rapidly.

The mechanical effects of a more coordinated contraction result in a shortening of the isovolumetric contraction phase and the pre-ejection time, and an increase in LV dP/dt (change in left ventricular pressure over time. The concept of measuring contractility with an implantable accelerometer was first clinically validated through a multicenter study on a rate responsive pacing system (BEST - Living from SORIN Biomedica) in 1996. This study positively demonstrates that measurement of Peak Endocardial Acceleration signal (called PEA or SonR) is feasible and reliable in the long-term, both for the purpose of rate response and as a hemodynamic monitor of cardiac function.

More recent clinical studies have demonstrated that optimal VV and AV Delays determined using algorithms based on SonR signal analysis (SonR method) are correlated with the highest hemodynamic improvement and lead to significant clinical benefit for the patients, thus reducing the rate of non-responsiveness to CRT therapy.

Therefore, automatic AV and VV delay optimization in patients with CRT devices could benefit both the patient and physician.

ELIGIBILITY:
Inclusion Criteria:

1. Patient eligible with class I and IIa indication for implantation of a CRT-D device according to current available guidelines ;
2. Modere,Severe HF (NYHA Class III or ambulatory IV)
3. LVEF ≤ 35 %
4. LBBB: QRS ≥ 120 ms ; non-LBBB : QRS ≥ 150 ms
5. On a stable, optimal drug regimen
6. Patient is in sinus rhythm at the time of enrollment;
7. Signed and dated informed consent

Exclusion Criteria:

1. Ventricular tachyarrhythmia of transient or reversible causes such as acute myocardial infarction, digitalis intoxication, drowning, electrocution, electrolyte imbalance, hypoxia or sepsis, uncorrected at the time of the enrolment;
2. Incessant ventricular tachyarrhythmia;
3. Unstable angina, or acute MI, CABG, or PTCA within the past 4 weeks;
4. Correctable valvular disease that is the primary cause of heart failure;
5. Recent CVA or TIA (within the previous 3 months);
6. Persistent or permanent atrial arrhythmias (or cardioversion for atrial fibrillation) within the past month;
7. Post heart transplant (patients who are waiting for a heart transplant are allowed in the study);
8. Renal failure (GFR<15 ml/min/1.73m2) or on dialysis
9. Previous implant with a CRT/CRT-D device;
10. Concurrent implant with another pacemaker or ICD (previously implanted pacemaker or ICD devices or RA leads should be removed prior to implant with the Paradym RF SONR CRT-D);
11. Already included in another clinical study that could confound the results of this study;
12. Life expectancy less than 1 year;
13. Inability to understand the purpose of the study or to understand and complete the QOL questionnaire;
14. Unavailability for scheduled follow-up or refusal to cooperate;
15. Sensitivity to 1 mg dexamethasone sodium phosphate (DSP)
16. Age of less than 18 years;
17. Pregnancy
18. Drug addiction or abuse
19. Under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1039 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of SonR CRT Optimization Effectiveness in terms of proportion of responders at 12 months. The investigational(SonR)and control groups(ECHO)will be compared in a non-inferiority context employing a clinically meaningful difference of 10%. | 12 months
  The analysis will be done on all patients implanted with the entire system who have been followed out to 12 months. The patients will be classified as improved, unchanged or worsened based on composite criteria(death/heart failure (HF) events,New York Heart association(NYHA) class), Quality of life (QOL).
  In the event that the non-inferiority test is met, a test of superiority will be conducted comparing the treatment and control groups.
Evaluation of Lead Safety: Acute SonRTipLead Complication-Free Rate (at 3 months) | 3 months
  SonRtip acute lead-related complication-free rate is defined as the proportion of patients not experiencing any complication related to the SonRtip lead within 3 months post-implant, relative to the total number of patients implanted with the lead.All patients who are successfully implanted with SonRtip lead will be included.
Evaluation of Lead Safety: Chronic SonRTipLead Complication-Free Rate (from 3 months to 12 months) | 12 months
  SonRtip lead-related complication-free rate is defined as the proportion of patients not experiencing any complication related to the SonRtip lead from 3 to 12 months post-implant.All patients who are successfully implanted with SonRtip lead will be included.

SECONDARY OUTCOMES:
Evaluation of CRT effectiveness and CRT Safety: evaluation of Mortality and HF hospitalizations at 12 months | 12 months
  This endpoint will compare treatment arms in a non-inferiority hypothesis test of the proportion of subjects that either died from any cause, or were hospitalized for heart failure
Evaluation of CRT effectiveness and CRT therapy: Proportion of patients worsened at 12 months | 12 months
  This endpoint will compare treatment arms in a non-inferiority hypothesis test of the proportion of subjects classified as worsened, in order to evaluate the potential detrimental effects of the optimization method
SonR tip lead pacing threshold | 24 months
  For all patients implanted with the SonRtip lead.
SonR tip lead sensing threshold | 24 months
  For all patients implanted with the SonRtip lead.
SonR tip lead pacing impedance | 24 months
  For all patients implanted with the SonRtip lead.
Evaluation of CRT effectiveness and CRT and System Safety: Report deaths for any cause | 24 months
  The report of the deaths occurred consists of the percentage of dead patients, the causes of death, the time to death, the survival curves.
Report Heart Failure-related events to assess CRT effectiveness | 24 months
  For all patients implanted it will be reported the percentage of patients with events, number of events for patients, event type, time to first occurence, survival curves)
Report Quality of life (QOL) improvement to assess CRT effectiveness (percentage of patients with improvements in QOL) | 24 months
  In all patients implanted the evaluation of the Quality of Life Score will consist of reporting the percentage of patients who showed improvement in their KCCQ Score at each follow-up post-implant
Report NYHA class improvement to assess CRT effectiveness (the percentage of patients with improved in NYHA class) | 24 months
  In all patients implanted the evaluation of the NYHA Classification will consist of reporting the percentage of patients who improved at least one NYHA class at each follow-up post-implant
Evaluation of CRT effectiveness: Report echocardiographic parameters trend at M12 | 12 months
  The intra-patient variations of the echocardiographic parameters measured at M12 as compared to those measured at baseline. The echo measures will be validated by an independent and blinded core lab
Evaluation of SonR CRT Optimization Effectiveness - Superiority by assessment the proportion of responder patients in SonR group | 18/24 months
  The analysis will be done on all patients implanted with the entire system. The patients will be classified as improved, unchanged or worsened based on composite criteria(death/heart failure events,NYHA class, Quality of life (QOL).
Evaluation of the time spent for CRT optimization by the physician on optimization in each group (sonR and ECHO) | 24 months
  The amount of time (mean, median, standard deviation, minimum, maximum)in each group will be evaluated in all patients implanted
Evaluation of the Number of re-optimizations performed in both groups (SonR and ECHO) | 24 months
  In all patients implanted will be evaluated the number of re-optimizations performed (mean, median, standard deviation, minimum, maximum) in each group (study and control).
Report Adverse Events for both group to assess CRT effectiveness / System Safety | 24 months
  For all patients enrolled all Adverse Events will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Brugada, Principal Investigator — Hospital Clinic of Barcelona
Locations (125):
- United States (31):
  - Brookwood Medical Center CardioVascular Associates, Birmingham, Alabama
  - AZ Heart Rhythm Center, Phoenix, Arizona
  - Brotman Medical Center, Culver City, California
  - Hoag Hospital, Newport Beach, California
  - Scripps Mercy Hospital, San Diego, California
  - Broward General Medical Center, Fort Lauderdale, Florida
  - St. Vincent's HealthCare, Jacksonville, Florida
  - Piedmont Hospital Research Institute, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - The University of Chicago Medicine Hospital, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital-CAS, Boston, Massachusetts
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - St. Luke's Roosevelt Hospital Center, New York, New York
  - New York Presbyterian, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Forsyth Hospital, Winston-Salem, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - St. Francis Hospital, Tulsa, Oklahoma
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Hospital of the University of PA, Philadelphia, Pennsylvania
  - Lexington Cardiology, Columbia, South Carolina
  - Providence Cardiology d/b/a South Caroline Heart Center, Columbia, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - VA North Texas Health Care System, Dallas, Texas
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - Plaza Medical Center of Fort Worth, Fort Worth, Texas
- Australia (2):
  - Princess Alexandra Hospital, Brisbane
  - Royal Perth Hospital, Perth
- Austria (5):
  - LKH Feldkirch, Feldkirch
  - Lkh Innsbruck - Invasoren Kardiologie - Innere Medizin, Innsbruck
  - KH Hietzing,4. Medizinische Abteilung Mit Kardiologie, Vienna
  - Wilhelminenspital, Vienna
  - SMZ-Ost, 1 Medizinische Abteilung, Vienna
- France (15):
  - Hôpital de la Cavale Blanche-CHU BREST, Brest
  - CHU - Hopital Michallon, Grenoble
  - CHRU de Lille,Hôpital Cardiologique, Lille
  - Centre Hospitalier Universitaire de La Timone, Marseille
  - Institut Jacques Cartier, Massy
  - Nouvelles Cliniques Nantaises, Nantes
  - InParys CLINIQUE BIZET, Paris
  - CHU de Bordeaux, Groupe hospitalier Sud, Hôpital Haut-L'évêque, Pessac
  - CH Poitiers, Poitiers
  - CHU Charles Nicolle, Rouen
  - CHU - Hopital Nord, Saint-Etienne
  - CH de Rangueil, Toulouse
  - Chru Trousseau, Tours
  - CHU Brabois, Vandœuvre-lès-Nancy
  - La Clinique du Tonkin, Villeurbanne
- Germany (17):
  - Herz- und Gefässzentrum Bad Bevensen, Bad Bevensen
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - St.-Marien-Hospital, Bonn
  - Universitätskliniken Bonn, Bonn
  - Klinikum Coburg, Coburg
  - Kardiocentrum Frankfurt and der Klinik Rotes Kreuz, Frankfurt
  - Universitäts-Herzzentrum Freiburg, Freiburg im Breisgau
  - Albertinen-Krankenhaus, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Schleswig-HolsteinCampus Kiel, Kiel
  - Klinikum Ludwigshafen, Ludwigshafen
  - Klinikum Magdeburg gemeinnützige GmbH, Magdeburg
  - Klinikum Grosshadern, München
  - Universitätsklinik Münster Innere Medizin C, Münster
  - Krankenhaus Reinbek St. Adolf-Stift, Reinbek
- Italy (20):
  - Ospedale Civile Ss. Antonio E Biago, Alessandria
  - Az. Osp-Univ. Ospedali Riuniti Umberto I-Lancisi-Salesi, Ancona
  - Azienda Ospedaliera S. Anna e S. Sebastiano, Caserta
  - AOU Ferrarotti-Alessi, Catania
  - Ospedale Maurizio Bufalini, Cesena
  - Azienda Ospedaliera S. Croce E Carle, Cuneo
  - Azienda Osped-Universitaria CAREGGI, Florence
  - Casa Di Cura Montevergine, Mercogliano
  - Osp. Niguarda, Milan
  - Ospedale Civile, Mirano
  - SUN Ospedale Monaldi, Napoli
  - Fondazione Toscana Gabriele Monasterio, Pisa
  - Policlinico Casilino, Roma
  - Osp. S. Maria della Misericordia, Rovigo
  - IRCCS Multimedica, Sesto San Giovanni
  - A.O. Città della Salute e della Scienza di Torino Cardiologia 1 - U, Torino
  - A.O. Città della Salute e della Scienza di Torino Cardiologia 2 ospedaliera, Torino
  - Ospedale Cà Foncello, Treviso
  - Azienda Ospedaliero-Universitaria Ospedali Riuniti di Trieste, Trieste
  - Az. Osp. Univ. S. Maria della Misericordia, Udine
- Netherlands (6):
  - Slingeland Ziekenhuis, Doetinchem
  - Erasmus MC : University Medical Center, Rotterdam
  - Vlietland Ziekenhuis, Schiedam
  - Sint Elisabeth Ziekenhuis, Tilburg
  - Ziekenhuis Bernhoven, Veghel
  - ISALA Klinieken, Zwolle
- Portugal (5):
  - Hospital Professor Doutor Fernando Fonseca, Amadora
  - Centro Hospitalar Lisboa Ocidental -Hospital de Santa Cruz (CHLO), Carnaxide
  - Hospital Santa Maria, Lisbon
  - Centro Hospitalar do Porto CHP Hospital de Santo Antonio, Porto
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
- Klinični center Ljubljana, Ljubljana, Slovenia
- Spain (14):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinico de Barcelona, Barcelona
  - Hospital Donostia, Donostia / San Sebastian
  - H. Virgen de las Nieves, Granada
  - Hospital Universitario La Paz, Madrid
  - Hospital Puerta de Hierro, Majadahonda
  - Hospital Universitario Virgen de la Victoria, Málaga
  - H. Universitario Central de Asturias, Oviedo
  - Hospital Universitario Marques de Valdecilla Sur, Santander
  - Hospital Virgen de Valme, Seville
  - H. General Universit., Valencia
  - CHU VIGO, Vigo
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois Lausanne (CHUV), Lausanne
  - Fondazione Cardiocentro Ticino, Lugano
- United Kingdom (7):
  - Queen Elizabeth Hospital, Birmingham
  - Papworth Everard, Cambridge
  - Ashford and St. Peter's Hospitals NHS Trust, Chertsey
  - Castle Hill Hospital Hull and East Yorkshire Hospitals NHS T, Cottingham
  - Leeds General Infirmary, Leeds
  - Genfield General Hospital, Leicester
  - King's College Hospital NHS Foundation Trust, London

REFERENCES:
- [Derived] Brugada J, Delnoy PP, Brachmann J, Reynolds D, Padeletti L, Noelker G, Kantipudi C, Rubin Lopez JM, Dichtl W, Borri-Brunetto A, Verhees L, Ritter P, Singh JP; RESPOND CRT Investigators. Contractility sensor-guided optimization of cardiac resynchronization therapy: results from the RESPOND-CRT trial. Eur Heart J. 2017 Mar 7;38(10):730-738. doi: 10.1093/eurheartj/ehw526. PMID 27941020
- [Derived] Brugada J, Brachmann J, Delnoy PP, Padeletti L, Reynolds D, Ritter P, Borri-Brunetto A, Singh JP. Automatic optimization of cardiac resynchronization therapy using SonR-rationale and design of the clinical trial of the SonRtip lead and automatic AV-VV optimization algorithm in the paradym RF SonR CRT-D (RESPOND CRT) trial. Am Heart J. 2014 Apr;167(4):429-36. doi: 10.1016/j.ahj.2013.12.007. Epub 2013 Dec 19. PMID 24655689